CLINICAL TRIAL: NCT01935817
Title: Silybin - Vitamin E- Phospholipids Complex Reduces Liver Fibrosis in Patients With Chronic Hepatitis C Treated With Peg-IFN-a and RBV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, A.P., University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: unict11/1997
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Silybin; Vitamin E; Phospholipids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Silybin + vitamin E + phospholipids complex (Active Comparator): Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg in one pill per day for 12 months
  Interventions: Drug: Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg complex
- sugar pill (Placebo Comparator): one placebo pill per day for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg complex
  Arms: Silybin + vitamin E + phospholipids complex
Drug: Placebo
  Arms: sugar pill

SUMMARY:
Chronic hepatitis C is both a virologic and a fibrotic disease, with mortality resulting mainly from the complications of cirrhosis and HCC.

The investigators' aim will be to evaluate the impact on of supplementation with a new pharmaceutical complex of silybin-vitamin E-phospholipids in patients with chronic hepatitis C treated with Pegylated-Interferon-α2b plus Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* infection by HCV
* under treatment with pegylated interferon 2 alpha and ribavirin

Exclusion Criteria:

* other liver diseases
* cancer
* severe jaundice
* pulmonary and renal chronic diseases
* prostatic diseases
* autoimmune diseases
* diabetes mellitus

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
transforming growth factor beta | 12 months
  serum marker of liver fibrosis

SECONDARY OUTCOMES:
hyaluronic acid | 12 months
  serum marker of liver fibrosis

OTHER OUTCOMES:
metalloproteinase 2 | 12 months
  serum marker of liver fibrosis
amino-terminal pro-peptide of type III procollagen | 12 months
  serum marker of liver fibrosis
tissue inhibitor of matrix metalloproteinase type I | 12 months
  serum marker of liver fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cannizzaro Hospital, Catania, Sicily, Italy